CLINICAL TRIAL: NCT00775346
Title: A Multi-Center Study to Assess the Performance of the Saturation Pattern Detection (SPD) Software Algorithm.
Brief Title: A Multi-Center Study to Assess the Performance of Saturation Patterns.
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 04212008; 20081155 (Other: Western Institutional Review Board)
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2010-06-16 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Sleep-Disordered Breathing; Obstructive Sleep Apnea; Sleep Apnea; Central Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Polysomnography (PSG) Subjects: Subjects who have been prescribed with needing a polysomnography (PSG) will be enrolled into the study.

SUMMARY:
A multi-center, prospective, single-visit study designed to acquire physiologic pulse oximeter waveform data during standard polysomnography (PSG) studies performed at multiple different Sleep Lab Centers.

DETAILED DESCRIPTION:
The polysomnograms are clinically indicated studies in patients suspected of having sleep-disordered breathing, including, but not limited to: obstructive sleep apnea, complex sleep apnea and/or central sleep apnea. Subjects who have been prescribed with needing a polysomnography (PSG) will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be referred to the Sleep Lab Center for evaluation of possible sleep-disordered breathing.
* Polysomnography (PSG) is obtained as part of normal, standard clinical practice.
* Subject is able to and willingly signs the informed consent form.

Exclusion Criteria:

* Subject and/or parent/legal guardian is, in the opinion of the investigator, mentally and/or physically unable to provide informed consent/child assent and/or to complete all requirements of the protocol.
* Subject is currently participating in or has participated in an investigational drug study within seven (7) days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are undergoing a standard sleep lab study/evaluation will have their data analyzed for this clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Mecca, MD, Study Chair — Medtronic - MITG
Locations (3):
- United States (3):
  - SleepFit, Broomfield, Colorado
  - Clayton Sleep Institute, Maplewood, Missouri
  - Sleep Medicine Centers, West Seneca, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 08/19/2008 to 10/14/2008 from 3 medical clinics in the United States.
Period: Overall Study
Arm/Group | Polysomnography (PSG) Subjects
Started | 92
Completed | 92
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Polysomnography (PSG) Subjects
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 51
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity Data of the Saturation Pattern Detection (SPD) Feature as a Predictor of Repetitive Reductions in Airflow (RRiA).
Description: Sensitivity and specificity were computed from the count of instances in which the Saturation Pattern Detection (SPD) index value (vs. Polysomnography) within a discrete ten minute interval correctly identified a Repetitive Reduction in Airflow (RRiA) as being present within that interval (True Positive), absent (True Negative), or incorrectly identified presence or absence (False Positive and False Negative, respectively). Sensitivity is True Positive divided by True Positive plus False Negative TP/(TP+FN). Specificity is True Positive divided by True Negative plus False Positive TP/(TN+FP).
Time Frame: 9 Hours
Measure: Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Polysomnography (PSG) Subjects
Number analyzed (Participants) | 92
Ratio
  Sensitivity of Automated Assessment | 0.820 [0.773 to 0.861]
  Specificity of Automated Assessment | 0.897 [0.883 to 0.910]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Polysomnography (PSG) Subjects
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other